CLINICAL TRIAL: NCT04824560
Title: Evaluating the Effect of an Evidence-Based One Page With Supplemental Visual Aids on the Knowledge and Perceptions of Blood Pressure Management Among Adults With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-458
Record Dates: First submitted 2021-03-09; First posted 2021-04-01 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BP Education (Other): All participants enrolled receive blood pressure education.
  Interventions: Behavioral: Blood pressure education

INTERVENTIONS:
Behavioral: Blood pressure education — One page teaching protocol performed by pharmacy students; phone follow-up

SUMMARY:
The purpose of this study is to evaluate changes in patient knowledge of blood pressure management and perceptions of making lifestyle changes to manage their blood pressure after implementation of an evidence-based one-page teaching protocol with supplemental handouts and optional use of suggested apps and web sites.

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 to 75 years old
* Ability to self-consent
* English-speaking
* Able to read/write English
* Currently prescribed at least one medication for treatment of essential primary hypertension

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Walgreens Store #6587, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BP Education
Started | 17
Completed | 5
Not Completed | 12

BASELINE CHARACTERISTICS:
Population: A total of 5 participants received the information, participated in follow-up phone calls, and returned all of their information in the provided SASE to the clinic.
Arm/Group | BP Education
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 54 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 3
  Race/Ethnicity: Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Pre & Post Survey & Knowledge Test
Description: change in participant's knowledge of blood pressure management as measured by a pre- and post-test of 10 multiple-choice questions
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: percentage of questions answered correct
Groups:
- BP Education: All participants enrolled receive blood pressure education; measured change in participant's knowledge of blood pressure management as measured by a pre- and post-test of 10 multiple-choice questions
Arm/Group | BP Education
Number analyzed (Participants) | 5
percentage of questions answered correct
  Pre-Test Knowledge Score | 85 [70 to 100]
  Post-Test Knowledge Score | 100 [100 to 100]

2. Secondary Outcome: BP Education Helpfulness
Description: All participants enrolled receive blood pressure education; measured patient's perceived helpfulness of educational one-page handout in a post-survey
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BP Education
Number analyzed (Participants) | 5
Participants
  Helpful - Yes | 4
  Helpful - NO | 1

3. Secondary Outcome: BP Education - Change in Confidence in Managing Disease State (Pre & Post Survey)
Description: change in participant's confidence in managing disease state as measured by pre & post survey
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BP Education
Number analyzed (Participants) | 5
Participants
  Pre-Survey: Confident in ability to manage disease state - pre-survey - Yes | 4
  Pre-Survey: Confident in ability to manage disease state - pre-survey - No | 1
  Post-Survey: Confident in ability to manage disease state - pre-survey - Yes | 4
  Post-Survey: Confident in ability to manage disease state - pre-survey - No | 1

ADVERSE EVENTS:
Time Frame: After enrollment, packet was mailed to participant and future phone call time frames set up to be able to call the participants back for an initial call to ensure packet received within one week of enrollment; with follow-up at 4 weeks after enrollment, 8 weeks after enrollment, and then a final phone call to ensure information would be mailed back at up to 4 weeks after the final phone call.
Description: As the intervention was a survey and phone call, no serious adverse events were expected and none were reported by participants within one week; 4 weeks, or 8 weeks,or when contacted to ensure information would be mailed back at up to 4 weeks after the final phone call (within a maximum of 12 weeks of enrollment).
Arm/Group | BP Education
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT04824560/Prot_SAP_001.pdf
  • Informed Consent Form (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT04824560/ICF_000.pdf